CLINICAL TRIAL: NCT03057418
Title: Open-label Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Auriхim Multiple Doses in Patients With Recurrent/Refractory В-cell, CD20-positive Non-Hodgkin Lymphoma of Low Tumor Grade or With Follicular Lymphoma
Brief Title: Open-label Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Auriхim
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biointegrator LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-CON4619-01
Record Dates: First submitted 2017-02-08; First posted 2017-02-20 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aurixim (Experimental): Dosage: 125 mg/m2, 250 mg/m2, 375 mg/m2 and 500 mg/m2. Formulation: concentrate for preparation of infusions 500 mg/50 ml and 100 mg/10 ml.
  Mode of administration: intravenous.
  Interventions: Drug: Aurixim

INTERVENTIONS:
Drug: Aurixim — Administration will be performed once a week during 4-week induction period, and then once per 12 weeks during supporting period, if necessary. Total maximum duration of the investigational therapy - 1 year, during which patients will receive up to 8 infusions of Aurixim.
  Other Names: CON-4619

SUMMARY:
This is an open-label study of safety, tolerability, pharmacokinetics and pharmacodynamics of Auriхim multiple doses in patients with recurrent/ refractory В-cell, CD20-positive non-Hodgkin lymphoma of low tumor grade or with follicular lymphoma, as well as in patients non-treated before for В-cell, CD20-positive non-Hodgkin lymphoma of low tumor grade.

The study will be carried out in 4-6 Russian and Belarussian sites. The study will be consisted of screening period, induction (obligatory) phase and supporting (non-obligatory) phase of the investigational therapy and post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

To participate in the clinical study, patients must comply to the following criteria:

1. Signed patient's information sheet and informed consent form
2. Males and females aged ≥ 18 years
3. The expected survival time not less than 6 months, with no need of an urgent intervention to eliminate life-threatening complications
4. Histologically and clinically confirmed at the screening diagnosis of В-cell, CD20-positive non-Hodgkin lymphoma of low tumor grade or follicular lymphoma, according to WHO's (World Health Organization) classification as of year 2008, namely:

   * Follicular lymphoma, cytological stage 1, 2 and 3a
   * Lymphoma from small lymphocytes (Small Lymphocytic Lymphoma) with number of peripheral blood lymphocytes < 5,000/mсl
   * Lymphoplasmacytic lymphoma, including Waldenstrom's macroglobulinemia with paraprotein meaning (IgM ) > 2,0 g/l
   * Extranodal marginal zone B-cell lymphoma of MALT-type
   * Nodal marginal zone B-cell lymphoma (± monocytoid В- lymphocytes)
   * Lymphoma of lien marginal zone cells.
5. Patients did not receive any therapy for the main disease, or disease recurrence, or refractivity after the previous therapy
6. II, III or IV disease stage according to Ann Arbor's classification and indications for immunotherapy, in the Investigator's opinion
7. The patient must have at least one 2-view measurable lesion (size by the long axis > 1,5 cm and size by the short axis > 1,0 cm, measured by means of CT scanner), that did not undergo radiotherapy in the past or appeared again in the course of the previous treatment.
8. Patients must have an ECOG status of 0 - 2
9. Requirements for laboratory parameters determined below:

   Hematology: Absolute neutrophil count:

   Platelets:

   Hemoglobin: ≥ 1500/mm3 (1.5 x 109 cells/L)
   * 100 000/mm3 (100 x 109 cells/L)
   * 8.0 g/dl

   Liver function: Total bilirubin:

   Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): ≤ 1.5 x ULN

   ≤ 2.5 x ULN Renal function: GFR (according to Cocroft-Golt formula): > 30 ml/min.
10. The patients must be practicing effective methods of birth control during the whole period of the study and 12 months after the last administration of the investigational product.

Exclusion Criteria:

The patient will be considered ineligible for the study in case he/she has any criteria listed here below:

1. Chronic lymphocytic leukemia
2. CNS invasion now or in the history (lymphoma of CNS or lymphomatous meningitis)
3. Treatment by chemotherapeutic agents or radiotherapy within 4 weeks before screening, treatment by nitrosourea and mitomycin C within 6 weeks before screening or presence of ongoing toxicities of ≥ II grade according to CTCAE, related to the prior therapy (excluding alopecia)
4. Prior treatment by MAb (monoclonal antibodies) within 3 months before screening
5. Concomitant immunosupressive therapy and systemic treatment by corticosteroids on the moment of screening.
6. Clinically significant cardiovascular diseases:

   * Myocardial infarction within 6 months before screening
   * Unstable angina within 3 months before screening
   * Congestive heart failure Class III or IV according to the New York Heart Association (NYHA) criteria
   * Clinically significant ventricular arrhythmia (ventricular tachycardia, ventricular fibrillation)
   * QTc interval > 460 ms (ECG) (calculated according to Fredericia formula), or a diagnosis of long QTc syndrome
   * Ejection fraction of left ventricle ≤ 50% (EchoCG)
   * Hypotension (systolic arterial blood pressure < 86 mm of mercury) or bradycardia with a heart rate of < 50 beats per min., except when caused by medications (e.g. beta-blockers)
   * Uncontrolled arterial hypertension (systolic arterial blood pressure > 170 mm of mercury or diastolic arterial blood pressure > 105 mm of mercury)
7. Peripheral neuropathy ≥ III severity level
8. Primary or secondary immunodeficiency now or in the history
9. Presence of antibodies to human immunodeficiency virus (HIV), or hepatitis С virus (HCV), active hepatitis B
10. Tuberculosis during last 5 years or positive result of the Quantiferon test
11. Active infection within 4 weeks before screening
12. Surgical interference (excluding biopsy of lymphatic nodes) within 4 weeks before screening
13. History of other malignancies with the exception of cervical carcinoma in situ or skin basal-cell carcinoma, that had undergone surgical removal and treatment within ≥ 5 years before screening
14. Uncontrolled concomitant diseases and conditions, including mental or social, which, in the Investigator's opinion, may prevent the patient from participation in the study.
15. Hypersensitivity to any of medicinal agents used in this study, to their compounds or to murine proteins, as well as significant, in the Investigator's opinion, allergic reactions in the history
16. Participation in other clinical studies or administration of other investigational products within 30 days before screening, or ongoing adverse reactions to any investigational product
17. Drug or alcohol abuse on the moment of screening or in the past, which, in the Investigator's opinion, makes the patient unsuitable for participation in the study.
18. Pregnant or lactating women, or women who plan to get pregnant during the clinical study; women of childbearing potential (not sterile and in postmenopause less than 2 years) who do not practice effective methods of birth control. Effective methods of birth control include usage of:

    * oral, injectable or transdermal contraceptives
    * a condom or diaphragm (barrier method) with spermicide, or
    * intrauterine device
19. Inability to read or write, unwillingness to understand and comply with the procedures of the study protocol, as well as any other concomitant medical or serious mental conditions, that make the patient unsuitable for participation in the clinical study, limit the validity of informed consent receipt or may affect the patient's ability to participate in the study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Up to 24 weeks after the last dose
  The number of patients with treatment-related AEs assessed by CTCAE, abnormal laboratory values and instrumental tests (ECG) that are related to treatment.
Maximum tolerated dose (MTD) of Aurixim | at Day 36 after the first dose
  MTD is defined as maximum dose at which DLT occurs in more than 1 patient of 6

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Up to week 71
  PK analysis of multiple doses of Aurixim after single and multiple dosage
CD19+ | Up to week 71
  Pharmacodynamics (PD) of multiple doses of Aurixim after single and multiple
Peak Plasma Concentration (Cmax) | Up to week 71
  PK analysis of multiple doses of Aurixim after single and multiple dosage
Elimination half-life (T1/2) | Up to week 71
  PK analysis of multiple doses of Aurixim after single and multiple dosage

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - State Budgetary Public Healthcare Institution of the Nizhni Novgorod Region "Hospital of Ambulance of Dzerzhinsk city", Dzerzhinsk
  - Federal State Budgetary Institution "National Medical-Surgical Center n.a. N.I.Pirogov" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Institution "Russian Oncological Scientific Center n.a. N.N.Blokhin" of the Russian Academy of Medical Sciences, Moscow

IPD SHARING:
Plan to Share IPD: No